CLINICAL TRIAL: NCT01516346
Title: Effect of Organic Nitrates and Hydralazine on Wave Reflections and Left Ventricular Structure and Function in Heart Failure With Preserved Ejection Fraction
Brief Title: Vasodilator Therapy for Heart Failure and Preserved Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Julio A.Chirinos, Director of non-invasive imaging and Assistant Professor of Medicine, Corporal Michael J. Crescenz VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01340; 5R21AG043802-02 (NIH)
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure; Congestive Heart Failure
Keywords: Heart Failure; Heart failure with preserved ejection fraction (HFpEF); Vasodilators; Isosorbide dinitrate; Hydralazine; wave reflections; arterial stiffness; hemodynamics
MeSH Terms: conditions — Heart Failure | interventions — Isosorbide Dinitrate; Hydralazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Isosorbide dinitrate (Active Comparator): Research pharmacy-formulated capsules will be given to the subjects in two bottles. For this interventional arm, one of the bottles will contain the active ingredient Isosorbide Dinitrate and the other will contain placebo capsules.
  Dosage of Isosorbide Dinitrate will be 20mg (if Stage 1) OR 40mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing, if they tolerate Stage 1 dosing. Frequency is three times daily to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Interventions: Drug: Isosorbide Dinitrate
- Isosorbide dinitrate + Hydralazine (Active Comparator): Research pharmacy-formulated capsules will be given to the subjects in two bottles. For this interventional arm, one of the bottles will contain the active ingredient Isosorbide Dinitrate and the other will contain the active ingredient Hydralazine.
  Dosage of Isosorbide Dinitrate will be 20mg (if Stage 1) OR 40mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing, if they tolerate Stage 1 dosing. Frequency is three times daily to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Dosage of Hydralazine will be 37.5mg (if Stage 1) OR 75mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing, if they tolerate Stage 1 dosing. Frequency is three times daily, to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Interventions: Drug: Isosorbide Dinitrate + Hydralazine
- Placebo (Placebo Comparator): Research pharmacy-formulated capsules will be given to subjects in two bottles. For this interventional arm, both the bottles will contain placebo capsules.
  Dosage will be same regardless of up-titration from Stage 1 dosing to Stage 2 dosing. Frequency is three times daily, to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isosorbide Dinitrate — Enrolled subjects will be randomized in a blinded fashion to 1 isosorbide dinitrate capsule TID + 1 placebo capsule TID. In addition, all subjects will receive a single in-lab dose of 0.4 mg of sublingual nitroglycerine (open label) before randomization to the blinded study drugs. Subjects receiving isosorbide dinitrate will be given 20mg PO q8am, 2pm, and 8pm and will be titrated up to 40mg PO q8am, 2pm, and 8pm.
  Arms: Isosorbide dinitrate
Drug: Isosorbide Dinitrate + Hydralazine — Enrolled subjects will be randomized in a blinded fashion to 1 isosorbide dinitrate capsule TID + 1 hydralazine capsule TID. In addition, all subjects will receive a single in-lab dose of 0.4 mg of sublingual nitroglycerine (open label) before randomization to the blinded study drugs. Subjects receiving isosorbide dinitrate will be given 20mg PO q8am, 2pm, and 8pm and will be titrated up to 40mg PO q8am, 2pm, and 8pm. Subjects receiving hydralazine will be given 37.5mg PO q8am, 2pm, and 8pm and will be titrated up to 75mg PO q8am, 2pm, and 8pm.
  Arms: Isosorbide dinitrate + Hydralazine
Drug: Placebo — Enrolled subjects will be randomized in a blinded fashion to 2 placebo capsules TID. In addition, all subjects will receive a single in-lab dose of 0.4 mg of sublingual nitroglycerine (open label) before randomization to the blinded study drugs.
  Arms: Placebo

SUMMARY:
The main objective is to test the effect of prolonged therapy (24 weeks) with isosorbide dinitrate ± hydralazine on arterial wave reflections (primary endpoint). Secondary endpoints include left ventricular (LV) mass, fibrosis and diastolic function) and exercise capacity (assessed via the 6-minute walk test) in patients with Heart Failure and Preserved Ejection Fraction (HFPEF). We will also test the hypothesis that the reduction in arterial wave reflections induced by vasoactive therapy will correlate with the improvement in exercise capacity, LV mass, fibrosis and diastolic function. Finally, we will assess whether the hemodynamic response to an acute dose of sublingual nitroglycerin (NTG) can predict the sustained changes in the reflected wave and other hemodynamic parameters in response to chronic vasodilator therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Previous clinical diagnosis of heart failure with current New York Heart Association Class II-IV symptoms.
2. LV ejection fraction >50% on a clinically indicated echocardiogram or ventriculogram within 12 months prior to consent, in the absence of a change in cardiovascular status, as assessed by the principal investigators.
3. Must have had at least one of the following within the 12 months prior to consent

   1. Hospitalization for decompensated HF
   2. Acute treatment for HF with intravenous loop diuretic or hemofiltration.
   3. Chronic treatment with a loop diuretic for control of HF symptoms.
   4. Chronic diastolic dysfunction on echocardiography as evidenced by left atrial enlargement or at least stage II diastolic dysfunction.
   5. Documentation of elevated NT-pro BNP levels or other natriuretic peptide marker (BNP, ANP) according to the laboratory and assay upper limit of normal in the previous year.
4. Stable medical therapy as defined by:

   1. No addition or removal of ACE, ARB, beta-blockers, or calcium channel blockers (CCBs) for 30 days.
   2. No change in dosage of ACE, ARBs, beta-blockers or CCBs of more than 100% for 30 days.
   3. No change in diuretic dose for 10 days.

Exclusion Criteria:

1. Rhythm other than sinus rhythm (i.e., atrial fibrillation).
2. Neuromuscular, orthopedic or other non-cardiac condition that prevents patient from walking in a hallway.
3. Non-cardiac condition limiting life expectancy to less than one year, per physician judgment.
4. Current or anticipated future need for nitrate therapy.
5. Valve disease (> mild aortic or mitral stenosis; > moderate aortic or mitral regurgitation).
6. Hypertrophic cardiomyopathy.
7. Known infiltrative or inflammatory myocardial disease (amyloid, sarcoid).
8. Pericardial disease.
9. Primary pulmonary arteriopathy.
10. Have experienced a myocardial infarction or unstable angina, or have undergone percutaneous transluminal coronary angiography (PTCA) or coronary artery bypass grafting (CABG) within 60 days prior to consent, or requires either PTCA or CABG at the time of consent.
11. Other clinically important causes of dyspnea such as morbid obesity or significant lung disease defined by clinical judgment or use of steroids or oxygen for lung disease.
12. Systolic blood pressure < 110 mmHg or > 180 mm Hg.
13. Diastolic blood pressure < 40 mmHg or > 100 mmHg.
14. Resting heart rate (HR) > 100 bpm.
15. A history of reduced ejection fraction (EF<50%).
16. Severe renal dysfunction (estimated GFR <30 ml/min/1.73m2 by modified MDRD equation) GFR (mL/min/1.73 m2) = 175 x (Scr)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if African American) (conventional units), which would impede the safe administration of gadolinium for MRI studies contrast.
17. Hemoglobin <10 g/dL.
18. Patients with known severe liver disease (AST > 3x normal, alkaline phosphatase or bilirubin > 2x normal).
19. Patients with a clinically indicated stress test demonstrating significant ischemia within a year of enrollment which was not followed by percutaneous or surgical revascularization.
20. Listed for cardiac transplantation.
21. Allergy to isosorbide dinitrate or hydralazine.
22. Current therapy with phosphodiesterase inhibitors, such as sildenafil, vardenafil or tadalafil, since the combination of nitrates and phosphodiesterase inhibitors can result in severe hypotension.
23. We will also exclude patients who are not suitable candidates for a cardiac MRI by virtue of having the following absolute or relative contraindications: (i) Central nervous system aneurysm clips; (ii) Implanted neural stimulators; (iii) Implanted cardiac pacemaker or defibrillator; (iv) Cochlear implant; (v) Ocular foreign body (e.g. metal shavings); (vi) Other implanted medical devices: (e.g. drug infusion ports); (vii) Insulin pump; (viii) Metal shrapnel or bullet; (ix) Claustrophobia; (x) Extreme obesity rendering the patient unable to fit into narrow-bore scanners; (xi) Unwillingness of the patient to undergo a cardiac MRI. All patients with metallic implants will be individually evaluated prior to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-02-05 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio A Chirinos, MD, PhD, Principal Investigator — Philadelphia VA Medical Center & University of Pennsylvania
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bhuiyan T, Maurer MS. Heart Failure with Preserved Ejection Fraction: Persistent Diagnosis, Therapeutic Enigma. Curr Cardiovasc Risk Rep. 2011 Oct;5(5):440-449. doi: 10.1007/s12170-011-0184-2. PMID 22081782
- [Background] Chirinos JA, Segers P. Noninvasive evaluation of left ventricular afterload: part 1: pressure and flow measurements and basic principles of wave conduction and reflection. Hypertension. 2010 Oct;56(4):555-62. doi: 10.1161/HYPERTENSIONAHA.110.157321. Epub 2010 Aug 23. PMID 20733089
- [Background] Chirinos JA, Segers P. Noninvasive evaluation of left ventricular afterload: part 2: arterial pressure-flow and pressure-volume relations in humans. Hypertension. 2010 Oct;56(4):563-70. doi: 10.1161/HYPERTENSIONAHA.110.157339. Epub 2010 Aug 23. PMID 20733088
- [Background] Endo H, Shiraishi H, Yanagisawa M. Afterload reduction by hydralazine in children with a ventricular septal defect as determined by aortic input impedance. Cardiovasc Drugs Ther. 1994 Feb;8(1):161-6. doi: 10.1007/BF00877105. PMID 8086327
- [Background] Greig LD, Leslie SJ, Gibb FW, Tan S, Newby DE, Webb DJ. Comparative effects of glyceryl trinitrate and amyl nitrite on pulse wave reflection and augmentation index. Br J Clin Pharmacol. 2005 Mar;59(3):265-70. doi: 10.1111/j.1365-2125.2004.02334.x. PMID 15752371
- [Background] Lind L, Pettersson K, Johansson K. Analysis of endothelium-dependent vasodilation by use of the radial artery pulse wave obtained by applanation tonometry. Clin Physiol Funct Imaging. 2003 Jan;23(1):50-7. doi: 10.1046/j.1475-097x.2003.00469.x. PMID 12558614
- [Background] Bradley JG, Davis KA. Orthostatic hypotension. Am Fam Physician. 2003 Dec 15;68(12):2393-8. PMID 14705758
- [Background] Downing GJ, Maulik D, Phillips C, Kadado TR. In vivo correlation of Doppler waveform analysis with arterial input impedance parameters. Ultrasound Med Biol. 1993;19(7):549-59. doi: 10.1016/0301-5629(93)90078-3. PMID 8310551
- [Background] Elkayam U, Bitar F. Effects of nitrates and hydralazine in heart failure: clinical evidence before the african american heart failure trial. Am J Cardiol. 2005 Oct 10;96(7B):37i-43i. doi: 10.1016/j.amjcard.2005.07.031. Epub 2005 Aug 9. PMID 16226934
- [Background] Brooks D, Solway S, Gibbons WJ. ATS statement on six-minute walk test. Am J Respir Crit Care Med. 2003 May 1;167(9):1287. doi: 10.1164/ajrccm.167.9.950. No abstract available. PMID 12714344
- [Derived] Chirinos JA, Bhattacharya P, Kumar A, Proto E, Konda P, Segers P, Akers SR, Townsend RR, Zamani P. Impact of Diabetes Mellitus on Ventricular Structure, Arterial Stiffness, and Pulsatile Hemodynamics in Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2019 Feb 19;8(4):e011457. doi: 10.1161/JAHA.118.011457. PMID 30764699
- [Derived] Zamani P, Akers S, Soto-Calderon H, Beraun M, Koppula MR, Varakantam S, Rawat D, Shiva-Kumar P, Haines PG, Chittams J, Townsend RR, Witschey WR, Segers P, Chirinos JA. Isosorbide Dinitrate, With or Without Hydralazine, Does Not Reduce Wave Reflections, Left Ventricular Hypertrophy, or Myocardial Fibrosis in Patients With Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2017 Feb 20;6(2):e004262. doi: 10.1161/JAHA.116.004262. PMID 28219917

RESULTS

PARTICIPANT FLOW:
Groups:
- Isosorbide Dinitrate: Dosage of Isosorbide Dinitrate will be 20mg (if Stage 1) OR 40mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing, if they tolerate Stage 1 dosing. Frequency is three times daily to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
- Isosorbide Dinitrate + Hydralazine: Dosage of Isosorbide Dinitrate will be 20mg (if Stage 1) OR 40mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing, if they tolerate Stage 1 dosing. Frequency is three times daily to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Dosage of Hydralazine will be 37.5mg (if Stage 1) OR 75mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing if they tolerate Stage 1 dosing. Frequency is three times daily, to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Isosorbide Dinitrate + Hydralazine: Enrolled subjects will be randomized in a blinded fashion to 1 isosorbide dinitrate capsule TID + 1 hydralazine capsule TID. In addition, all subjects will receive a single in-lab dose of 0.4 mg of sublingual nitroglycerine (open label) before randomization to the blinded study drugs. Subjects receiving isosorbide dinitrate will be given 20mg PO q8am, 2pm, and 8pm and will be titrated up to 40mg PO q8am, 2pm, and 8pm.
Period: Overall Study
Arm/Group | Isosorbide Dinitrate | Isosorbide Dinitrate + Hydralazine | Placebo
Started | 13 | 15 | 16
Completed | 7 | 9 | 11
Not Completed | 6 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Isosorbide Dinitrate + Hydralazine: Dosage of Isosorbide Dinitrate will be 20mg (if Stage 1) OR 40mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing, if they tolerate Stage 1 dosing. Frequency is three times daily to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Dosage of Hydralazine will be 37.5mg (if Stage 1) OR 75mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing, if they tolerate Stage 1 dosing. Frequency is three times daily, to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Isosorbide Dinitrate + Hydralazine: Enrolled subjects will be randomized in a blinded fashion to 1 isosorbide dinitrate capsule TID + 1 hydralazine capsule TID. In addition, all subjects will receive a single in-lab dose of 0.4 mg of sublingual nitroglycerine (open label) before randomization to the blinded study drugs. Subjects receiving isosorbide dinitrate will be given 20mg PO q8am, 2pm, and 8pm and will be titrated up to 40mg PO q8am, 2pm, and 8pm.
- Total: Total of all reporting groups
Arm/Group | Isosorbide Dinitrate | Isosorbide Dinitrate + Hydralazine | Placebo | Total
Number analyzed (Participants) | 13 | 15 | 16 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [56 to 65] | 60 [55 to 66] | 66.5 [59.5 to 72] | 62 [59 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 13
  Male | 8 | 11 | 12 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 10 | 9 | 27
  White | 4 | 5 | 7 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 16 | 44

OUTCOME MEASURES:

1. Primary Outcome: Wave Reflection Magnitude
Description: The dimensionless ratio of backward (reflected) to forward wave amplitude. Higher values imply more wave reflection.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: dimensionless ratio
Arm/Group | Isosorbide Dinitrate | Isosorbide Dinitrate + Hydralazine | Placebo
Number analyzed (Participants) | 13 | 14 | 15
dimensionless ratio | 0.38 [0.33 to 0.43] | 0.44 [0.37 to 0.51] | 0.37 [0.31 to 0.43]

2. Secondary Outcome: LV Mass
Description: LV mass measured by MRI, in grams normalized to height in meters raised to the 1.7 power (m^1.7)
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: grams / meters ^1.7
Arm/Group | Isosorbide Dinitrate | Isosorbide Dinitrate + Hydralazine | Placebo
Number analyzed (Participants) | 7 | 8 | 11
grams / meters ^1.7 | 68.2 [60 to 76.3] | 66.2 [61.4 to 71.1] | 67.2 [62.8 to 71.5]

3. Secondary Outcome: Quality of Life (Kansas City Cardiomyopathy Questionnaire Score)
Description: Quality of life, assessed with the Kansas City cardiomyopathy questionnaire (overall summary score, which ranges from 0 to 100). Higher values imply better quality of life.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: Points on a scale
Arm/Group | Isosorbide Dinitrate | Isosorbide Dinitrate + Hydralazine | Placebo
Number analyzed (Participants) | 11 | 13 | 16
Points on a scale | 62.1 [51.1 to 73.1] | 44.9 [37.1 to 62.7] | 62.1 [50.8 to 73.1]

4. Secondary Outcome: Early Diastolic Mitral Annular Velocity
Description: Diastolic mitral annular velocity measured at the basal septal mitral annulus
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: cm/s
Arm/Group | Isosorbide Dinitrate | Isosorbide Dinitrate + Hydralazine | Placebo
Number analyzed (Participants) | 13 | 15 | 15
cm/s | 6.8 [5.5 to 8.0] | 7.3 [6.1 to 8.6] | 6.5 [5.4 to 7.6]

5. Secondary Outcome: Myocardial Extracellular Volume Fraction
Description: Myocardial extracellular volume, expressed as percent of total tissue volume, measured by MRI (T1 mapping pre and post-gadolinium administration)
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Isosorbide Dinitrate | Isosorbide Dinitrate + Hydralazine | Placebo
Number analyzed (Participants) | 7 | 8 | 11
Percentage | 29.0 [25.0 to 33.0] | 31.3 [29.2 to 33.4] | 29.5 [26.4 to 32.6]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: None of the participants experienced mortality throughout the study.
Groups:
- Isosorbide Dinitrate: Research pharmacy-formulated capsules will be given to the subjects in two bottles. For this interventional arm, one of the bottles will contain the active ingredient Isosorbide Dinitrate and the other will contain placebo capsules.
  Dosage of Isosorbide Dinitrate will be 20mg (if Stage 1) OR 40mg (if Stage 2). All the subjects will be uptitrated to Stage 2 dosing, if they tolerate Stage 1 dosing. Frequency is three times daily to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Isosorbide Dinitrate: Enrolled subjects will be randomized in a blinded fashion to 1 isosorbide dinitrate capsule TID + 1 placebo capsule TID. In addition, all subjects will receive a single in-lab dose of 0.4 mg of sublingual nitroglycerine (open label) before randomization to the blinded study drugs. Subjects receiving isosorbide dinitrate will be given 20mg PO q8am, 2pm, and 8pm and will be titrated up to 40mg PO q8am, 2pm, and 8pm.
- Placebo: Research pharmacy-formulated capsules will be given to subjects in two bottles. For this interventional arm, both the bottles will contain placebo capsules.
  Dosage will be same regardless of up-titration from Stage 1 dosing to Stage 2 dosing. Frequency is three times daily, to be taken at 8 AM, 2 PM and 8 PM. Duration is for 24 weeks.
  Placebo: Enrolled subjects will be randomized in a blinded fashion to 2 placebo capsules TID. In addition, all subjects will receive a single in-lab dose of 0.4 mg of sublingual nitroglycerine (open label) before randomization to the blinded study drugs.
Arm/Group | Isosorbide Dinitrate | Isosorbide Dinitrate + Hydralazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 3/13 | 3/15 | 1/16
Other Adverse Events (participants affected / at risk) | 8/13 | 9/15 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isosorbide Dinitrate (N=13) | Isosorbide Dinitrate + Hydralazine (N=15) | Placebo (N=16)
Hospital Admission (Investigations) | 3 (4) | 3 (3) | 1 (3) — Admission to emergency room and/or hospital
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isosorbide Dinitrate (N=13) | Isosorbide Dinitrate + Hydralazine (N=15) | Placebo (N=16)
Headache (General disorders) | 4 (4) | 2 (2) | 1 (1)
GI Symptoms (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness/Lightheadedness (General disorders) | 2 (2) | 2 (2) | 0 (0)
Hypotension (General disorders) | 1 (1) | 3 (3) | 0 (0)
Orthostasis (General disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No